CLINICAL TRIAL: NCT00367120
Title: A Multicenter, Randomized, Open Label Comparative Study Of Azithromycin Extended Release (ZMAX) Versus Amoxicillin/Clavulanate Potassium In Subjects With Acute Bacterial Sinusitis (ABS) In A Physician Practice Environment
Brief Title: Zmax Compared to Augmentin in Sinusitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0661180
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Amoxicillin-Potassium Clavulanate Combination

INTERVENTIONS:
Drug: Azithromycin Extended Release
Drug: Amoxicillin/Clavulanate

SUMMARY:
This study will enroll patients with Bacterial Sinusitis who will be treated with either Zmax (Azithromycin Extended Release) or Augmentin (Amoxicillin/Clavulanate). The purpose of the study is to compare early resolution of symptoms between the two treatments. Patients will report resolution of their sinusitis symptoms through a daily questionnaire. There will be two follow-up telephone interviews on days 12 and 28 to evaluate quality of life, satisfaction with therapy, and use of healthcare services.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of acute uncomplicated bacterial maxillary sinusitis as demonstrated by presence of the following cardinal signs and symptoms for a minimum duration of 7 days, and no longer than 30 days:
* Facial pain, pressure and/or tightness over one or both maxillary sinuses, and/or pain in one or both maxillary areas that worsens with movement or percussion, and
* Presence of one or more of the following signs:
* Discolored (yellow-green) nasal discharge
* Discolored (yellow-green) drainage in the posterior pharynx
* Discolored (yellow-green) discharge from the maxillary sinus orifice
* Two or more of the following symptoms are present:
* Fever, as defined by:
* Oral temperature: >38C or >100.4F, or
* Tympanic temperature: >38.5C or >101.2F
* Frequent coughing
* Nasal congestion,
* Post-nasal drainage.

Exclusion Criteria:

* Treatment with any systemic antibiotic within 30 days prior to enrollment
* Symptoms of sinusitis lasting for longer than 30 days;
* Four or more episodes of acute sinusitis within the preceding 12 months;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 762 (Actual)
Dates: Start 2006-06; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Patient reported symptom resolution at day 5

SECONDARY OUTCOMES:
Time to symptom resolution.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661180&StudyName=Zmax+Compared+to+Augmentin+in+Sinusitis